CLINICAL TRIAL: NCT05043428
Title: The Roles of Peers and Functional Tasks in Enhancing Exercise Training for Adults With COPD: a Pilot Randomized Controlled Trial
Brief Title: The Roles of Peers and Functional Tasks in Enhancing Exercise Training for Adults With COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Fondation Québécoise en Santé Respiratoire (Unknown)
Responsible Party: Principal Investigator, Shane Norman Sweet, Associate Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 250965
Record Dates: First submitted 2021-08-27; First posted 2021-09-14 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: exercise; peer support; behavior change
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Intervention Model Description: A convenience sample of adults living with COPD (N=22) will be recruited to participate in an 8-week online exercise intervention. The objective is to test a two-arm pilot randomized controlled trial (RCT) for individuals living with COPD and to determine whether the intervention can improve individuals' performance in activities of daily and social living.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Those randomized to the intervention group will be asked to attend 16 online sessions (2 session/week). Each session will last one hour (total time: 16 hours. The exercise portion will be approximately 30 minutes of each session and led by a certified kinesiologist. These exercises are based on activities related to your daily life. As well, they will take part in peer support sessions. The peer support session will be approximately 30 minutes and be moderated by a behaviour change specialist who will also provide strategies to be active. In this peer support group, particpants will share and learn from other individuals living with COPD to help you stay active during and after the intervention. The online sessions will be video recorded to make sure that the program is delivered as designed.
  Interventions: Behavioral: The roles of peers and functional tasks in enhancing exercise training for adults with COPD: a pilot randomized controlled trial
- Control Group (Active Comparator): Those randomized to the control group will be asked to participate in an 8-week exercise program based on the exercise component of a standard home-based pulmonary rehabilitation program. During week 1 of the program, participants will receive a videocall via Microsoft Teams from the certified kinesiologist who will prescribe an exercise program, supervise the first exercise session, and provide a copy of Living Well with COPD, a list of strength exercises, and a home exercise diary. In weeks 2-8, participant exercises will be performed offline, on their own. Participants will be encouraged to engage in two or more exercise sessions per week, targeting both aerobic capacity and muscular strength, and document their exercise using a home diary. They will also receive a phone call once a week from the certified kinesiologist to discuss their exercise progress.
  Interventions: Behavioral: The roles of peers and functional tasks in enhancing exercise training for adults with COPD: a pilot randomized controlled trial

INTERVENTIONS:
Behavioral: The roles of peers and functional tasks in enhancing exercise training for adults with COPD: a pilot randomized controlled trial — An 8 week two-arm pilot randomized control trial aimed to evaluate the effects of an online exercise and peer support intervention for people living with COPD.

SUMMARY:
This study aims to evaluate the effects of an online exercise and peer support intervention for people living with COPD. In the framework of a randomized control trial, 24 adults with COPD will be recruited to participate in the study and will be randomly assigned to either the control or intervention group. The control group will participate in an 8-week virtual program based on the exercise component of a standard home-based pulmonary rehabilitation program (one online consultation and 7 phone calls with a kinesiologist). The intervention group will participate in a twice a week online intervention that includes an exercise component based on individuals' activities of daily living and a peer support component where individuals will be taught and encouraged to discuss behaviour change techniques that have been shown to help support increased participation in physical activity and/or exercise. The goal of this study is to determine the efficacy of the novel online exercise intervention and whether the benefits are above other intervention options.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be at least 18 years of age, have no diagnosed cognitive impairment, have a COPD diagnosis, be medically able to participate in exercise (confirmed by healthcare professional in the past 2 years), have access to a computer with a camera and internet, speak English or French, and have the intention to become physically active in the next 2 months or have been minimally active (<150 minutes per week) in the past 2 months

Exclusion Criteria:

* less than 18 years of age, diagnosed with a cognitive impairment, not diagnosed with COPD by a medical professional, unable to participate in exercise or unconfirmed in the past 2 years from a medical professional, no access to a computer and internet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Performance in activities of daily and social living | Baseline, 8 and 12 weeks
  Participant goal participation will be measured by improvement in initial goals set at the beginning of the study using the Canadian Occupation Performance Measures (COPM). Success will be determined by calculating individuals change score on their satisfaction with their performance in their target areas post-intervention. A change score of 2 on an item is said to represent significant change (Law et al., 2000). A change score of at least 2 on 50% of items (dependent on personal goals) for 70% of participants will be the indicator of success.

SECONDARY OUTCOMES:
Timed "Up & Go" test | Baseline, 8 and 12 weeks
  This test measures the time it takes an individual to stand from a standard chair (approximately 46cm), walk 3 metres, walk back, and return to sit on the chair (Podsiadlo & Richardson, 1991). The participant is timed from when the leave the seat to when they are seated again. A time of >30 seconds is the cut-off for safe unsupervised participation (Podsiadlo & Richardson, 1991). Anyone who gets a time >30seconds will be informed that they cannot participate.
1-minute sit-to-stand test | Baseline, 8 and 12 weeks
  The 1-minute sit-to-stand test is a measure of exercise capacity that has been validated with individuals living with COPD (Puhan et al., 2013). Individuals sit on a standard chair without arm rests, with their legs hip-width apart and about 90 degrees knee flexion and aligned and are asked to hold their hands stationary on their hips. Participants are then asked to stand and sit 1-2 times to familiar themselves with the movement. Then, for the duration of 1 minute, participants are asked to do as many repetitions as possible of the sit to stand, without using arms for support. The number of repetitions is recorded.
Handgrip Test | Baseline, 8 and 12 weeks
  To measure handgrip strength, we will use a Hand Dynamometer that will be sent to participants. Individuals sit with their shoulders adducted, elbows flexed to 90˚ and forearms in a neutral position (Puhan et al., 2013). They are then asked to squeeze the handle as much as possible and read to the nearest kilogram where the needle stopped, which is then recorded. The best of six measurements is used as an indication of upper body strength.
Borg Scale - Dyspnea | Baseline, 8 and 12 weeks
  On a scale from 0-10, participants' indicate their breathlessness level. 0- No breathlessness at all to 10- Maximal breathlessness
Godin Leisure Time Physical Activity Questionnaire | Baseline, 8, and 12 weeks
  Self-reported physical activity levels measured in length of bouts over the previous 7 days to determine physical activity frequency.
The Psychological Need Satisfaction in Exercise scale | Baseline, 8, and 12 weeks
  This 1-6 scale represents different feelings people have when they exercise. 1-true to how they typically feel when exercising, and 6-false to how they typically feel when exercising.
The Treatment Self-Regulation Questionnaire | Baseline, 8, and 12 weeks
  This 7 point scale relates to the reasons why one would either start to exercise regularly or continue to do so. 1- not at all true to the reason why they would exercise regularly, and 7- Very to true to the reason why they would exercise regularly.
Social Support from Peer Support Group Questionnaire | 8 and 12 weeks
  This 4 point scale measures how often during the past 4 weeks peers (i.e. other people with COPD) have provided informational and emotional support to the participant. 1- Never provided the support described and 4- Very often provided the support described.
Medical Research Council Questionnaire on Breathlessness (mMRC) | Baseline, 8, and 12 weeks
  This questionnaire was used to measure participants' breathlessness burden using a single item scale from 0 to 4, where a score of 0-1 indicated mild breathlessness and 2-4 indicated increased breathlessness.
COPD Assessment Test (CAT) | Baseline, 8, and 12 weeks
  This questionnaire was used to measure the impact COPD is having on well being and daily life. The CAT is an eight-item semantic differential scale from 0 to 5, where 0 is no impact and 5 is extremely impactful. Participants' scores were totaled and a score of ≥ 10 indicated higher than normal burden of disease.

OTHER OUTCOMES:
Activities, Healthcare, and Research Priorities Survey | Baseline, 8, and 12 weeks
  Participants will answer 26 questions based on daily and social activities and be asked if they participate in said activity. Responses include: Yes - as much as I want. Yes - but less than I want. No - but I would like to do it. No - and I don't want to do it.
Three Factor Social Identity Questionnaire | 8, and 12 weeks
  This 7 point scale measures feelings about being a part of the exercise and peer support group. 1-strongly disagree and 7- strongly agree to indicate agreement with each of the statements.
The Acceptability of Intervention Measure (AIM) | 8, and 12 weeks
  The Acceptability of Intervention Measure will be administered to measure high acceptability and satisfaction with the intervention. Using a 5 point scale, participants will answer 8 questions and rate them as 1- Completely disagree to 5- Completely agree.
Intervention Appropriateness Measure (IAM) | 8, and 12 weeks
  The Intervention Appropriateness Measure will be administered to measure high acceptability and satisfaction with the intervention. Using a 5 point scale, participants will answer 8 questions and rate them as 1- Completely disagree to 5- Completely agree.
Feasibility of Intervention Measure (FIM) | 8, and 12 weeks
  The Feasibility of Intervention Measure will be administered to measure high acceptability and satisfaction with the intervention. Using a 5 point scale, participants will answer 8 questions and rate them as 1- Completely disagree to 5- Completely agree.
6-Item Health Care Climate Questionnaire | 4, 8, and 12 weeks
  This 7 point scale measures how strongly the participant experienced interest, intrigue, focus, enjoyment, and annoyance during their participation in he Functional Tasks and Peer Support Intervention. 1-not at all experienced during the intervention to 7-extremely experienced during the intervention.
Behaviour Change Technique Usage Questionnaire | baseline, 8, and 12 weeks
  Participants completed a questionnaire that asked them to rate on a scale from 1 (not once) to 5 (daily) how frequently they have used goal setting, action planning, coping planning, physical restructuring, self monitoring, values identification, social restructuring, resource finding, and self belief in the past two weeks,

CONTACTS AND LOCATIONS:
Overall Officials: Shane Sweet, Ph.D, Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No